CLINICAL TRIAL: NCT00543855
Title: Double-blind Study of E2020 in Patients With Dementia With Lewy Bodies - Phase II
Brief Title: A Double-blind Study of E2020 (Donepezil Hydrochloride) in Patients With Dementia With Lewy Bodies (DLB) (Study E2020-J081-431)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-J081-431
Record Dates: First submitted 2007-10-04; First posted 2007-10-15 (Estimated); Results first posted 2013-02-18 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Dementia With Lewy Bodies (DLB)
Keywords: Lewy Body Disease; Dementia; Clinical Trial; Phase II; E2020; donepezil hydrochloride
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 3 mg Donepezil hydrochloride (Experimental)
  Interventions: Drug: 3 mg Donepezil hydrochloride
- 5 mg Donepezil hydrochloride (Experimental)
  Interventions: Drug: 5 mg Donepezil hydrochloride
- 10 mg Donepezil hydrochloride (Experimental)
  Interventions: Drug: 10 mg Donepezil hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 3 mg Donepezil hydrochloride — Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily for 12 weeks (Day 1- Day 84) after breakfast.
  Other Names: Aricept; Donepezil hydrochloride; E2020
  Arms: 3 mg Donepezil hydrochloride
Drug: 5 mg Donepezil hydrochloride — Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 1- Day 14 (2 weeks).
  Followed by one 5 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 15- Day 84 (10 weeks).
  Other Names: Aricept; Donepezil hydrochloride; E2020
  Arms: 5 mg Donepezil hydrochloride
Drug: 10 mg Donepezil hydrochloride — Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 1- Day 14 (2 weeks).
  Followed by one 5 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 15- Day 42 (4 weeks).
  Followed by two 5 mg Donepezil hydrochloride tablets (10 mg) by mouth, once daily after breakfast for Day 43 - Day 84 (6 weeks).
  Other Names: Aricept; Donepezil hydrochloride; E2020
  Arms: 10 mg Donepezil hydrochloride
Drug: Placebo — Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: Two Donepezil hydrochloride Placebo tablets by mouth, once daily for 12 weeks (Day 1- Day 84) after breakfast.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of E2020 in patients with Dementia with Lewy Bodies (DLB).

ELIGIBILITY:
Inclusion criteria:

Patients diagnosed as probable Dementia With Lewy Bodies (DLB) according to the diagnostic criteria for DLB.

Participants having caregivers who submit written consent for cooperative involvement in this study, can routinely stay with participants 3 days a week (at least 4 hours a day), provide participants' information necessary for this study, assist treatment compliance, and escort participants on required visits to study institution.

Exclusion criteria:

Participants with past experience of donepezil (Aricept) therapy at the same study institution.

Participants treated with donepezil in 3 months immediately before starting the observation period.

Participants with a complication of serious neuropsychiatric disease(s) such as stroke, brain tumor, schizophrenia, epilepsia, normal pressure hydrocephalus, mental retardation, brain trauma with unconsciousness, and/or experience of brain surgery causing unsolved deficiency.

Participants with severe complication of cardiovascular, hepatic, renal, hematological, or other diseases unable to secure the safety.

Pregnant or lactating women, or women who are willing to become pregnant no later than 1 month after the scheduled study completion

Participants with severe extrapyramidal disorders (Hoehn & Yahr staging score is ≥IV)

Participants whose systolic blood pressure is <90 mmHg or pulse rate is <50 beats/min.

Participants suspected to have a complication of vascular dementia based upon neurological findings.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2007-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masaki Nakagawa, Study Director — Neurosciences Clinical Development Section, Japan / Asia Clinical Research, Product Creation Unit, Eisai Product Creation System.
Locations (43):
- Japan (43):
  - Nagoya, Aichi-ken
  - Ōbu, Aichi-ken
  - Toyokawa, Aichi-ken
  - Akita, Akita
  - Chiba, Chiba
  - Fukui-shi, Fukui
  - Fukuoka, Fukuoka
  - Kurume, Fukuoka
  - Omuta, Fukuoka
  - Maebashi, Gunma
  - Miyoshi, Hiroshima
  - Ōtake, Hiroshima
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Tsukuba, Ibaraki
  - Kahoku, Ishikawa-ken
  - Morioka, Iwate
  - Yokohama, Kanagawa
  - Kochi, Kochi
  - Nankoku, Kochi
  - Kōshi, Kumamoto
  - Kumamoto, Kumamoto
  - Jōyō, Kyoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Komoro, Nagano
  - Kashihara, Nara
  - Jōetsu, Niigata
  - Sanjō, Niigata
  - Yufu, Oita Prefecture
  - Osaka, Osaka
  - Sakai, Osaka
  - Suita, Osaka
  - Saitama, Saitama
  - Izumo, Shimane
  - Shizuoka, Shizuoka
  - Bunkyo-ku, Tokyo
  - Kodaira, Tokyo
  - Koto-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Ube, Yamaguchi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 167 participants initiated the Observation period, 140 participants were enrolled in the treatment period, one participant did not receive treatment.
Groups:
- 3 mg Donepezil Hydrochloride: E2020 (Aricept) : Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily for 12 weeks (Day 1- Day 84) after breakfast.
- 5 mg Donepezil Hydrochloride: E2020 (Aricept) : Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 1- Day 14 (2 weeks).
  Followed by one 5 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 15- Day 84 (10 weeks).
- 10 mg Donepezil Hydrochloride: E2020 (Aricept) : Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 1- Day 14 (2 weeks).
  Followed by one 5 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 15- Day 42 (4 weeks).
  Followed by two 5 mg Donepezil hydrochloride tablets (10 mg) by mouth, once daily after breakfast for Day 43 - Day 84 (6 weeks).
- Placebo: Placebo : Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: Two Donepezil hydrochloride Placebo tablets by mouth, once daily for 12 weeks (Day 1- Day 84) after breakfast.
Period: Overall Study
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Started | 35 | 33 | 37 | 34
Completed | 31 | 31 | 31 | 30
Not Completed | 4 | 2 | 6 | 4
Not completed — Adverse Event | 3 | 1 | 3 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10 mg Donepezil Hydrochloride: E2020 (Aricept) : Observation Period: Two Donepezil hydrochloride placebo tablets once daily by mouth after breakfast for 2 weeks.
  Treatment Period: One 3 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 1- Day 14 (2 weeks).
  Followed by one 5 mg Donepezil hydrochloride tablet by mouth plus one Donepezil hydrochloride placebo tablet by mouth, once daily after breakfast for Day 15- Day 42 (4 weeks).
  Followed by two 5 mg Donepezil hydrochloride tablets (10 mg) by mouth, once daily after breakfast for Day 43- Day 84 (6 weeks).
- Total: Total of all reporting groups
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo | Total
Number analyzed (Participants) | 35 | 33 | 37 | 34 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 79.6 (4.5) | 77.9 (6.7) | 78.4 (6.1) | 78.7 (4.9) | 78.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 33 | 23 | 90
  Male | 17 | 17 | 4 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function: Change From Baseline in Mini-mental State Examination (MMSE) Total at Week 12 Last Observation Carried Forward (LOCF)
Description: MMSE measured general cognitive functioning: orientation, memory, attention, calculation, language, visuospatial functions. Total score derived from sub-scores; total ranged from 0 - 30, where a higher score indicated better cognitive state. Change: mean score at Week 12 LOCF minus mean score at baseline. Values at final evaluation were imputed using a Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline and every 4 weeks up to 12 weeks
Population: Per Protocol Set (PPS) was defined as those participants who complied with the study protocol.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Number analyzed (Participants) | 33 | 31 | 33 | 30
Score on a scale
  Baseline | 20.1 (4.2) | 19.7 (4.4) | 19.7 (4.5) | 18.2 (4.8)
  Change from Baseline (LOCF) | 1.2 (3.8) | 3.5 (3.2) | 2.3 (3.2) | -0.6 (2.7)

2. Primary Outcome: Psychiatric Symptoms: Change From Baseline in Neuropsychiatric Inventory (NPI) Total at Week 12 Last Observation Carried Forward (LOCF)
Description: NPI measured 10 different domains of psychiatric symptoms including delusion and hallucination. Each domain is scored for: present or absent, frequency, and severity. The score derived from sub-scores; total ranged from "0" to "120," higher score indicated "worse neuropsychiatric outcomes." Change: mean score at Week 12 LOCF minus mean score at baseline. Values at final evaluation were imputed using a Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline and every 4 weeks up to 12 weeks
Population: Per Protocol Set (PPS) was defined as those participants who complied with the study protocol.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Number analyzed (Participants) | 33 | 31 | 33 | 30
Score on a scale
  Baseline | 20.9 (13.1) | 14.2 (8.4) | 19.1 (11.8) | 18.4 (8.9)
  Change from Baseline (LOCF) | -4.3 (21.5) | -5.9 (6.5) | -10.2 (12.0) | -3.1 (10.9)

3. Primary Outcome: Global Clinical Function: Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC-plus) Total at Week 12 Last Observation Carried Forward (LOCF)
Description: CIBIC plus is a clinician's interview-based impression of change plus the caregiver's input. It is a seven-point categorical assessment scale for evaluating global clinical function, ranging from "markedly improved" to "markedly worse". Percentage of participants in each category were reported. Values at final evaluation were imputed using a Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline and week 12
Population: Per Protocol Set (PPS) was defined as those participants who complied with the study protocol.
Measure: Number; unit: Percentage of Participants
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Number analyzed (Participants) | 33 | 31 | 33 | 30
Percentage of Participants
  Marked improvement | 3.6 | 17.9 | 3.8 | 0
  Moderate Improvement | 17.9 | 17.9 | 11.5 | 3.7
  Minimal Improvement | 50.0 | 35.7 | 50.0 | 29.6
  No Change | 21.4 | 14.3 | 30.8 | 18.5
  Minimal Worsening | 3.6 | 7.1 | 3.8 | 37.0
  Moderate Worsening | 0 | 7.1 | 0 | 11.1
  Marked Worsening | 3.6 | 0 | 0 | 0

4. Primary Outcome: Burden on Caregiver: Change From Baseline in J-ZBI (Japanese- Zarit Caregiver Burden Interview) Total at Week 12 Last Observation Carried Forward (LOCF)
Description: J-ZBI is a Japanese version instrument to measure and assess the level of burden experienced by the principal caregivers of participants with dementia.
  ZBI contains 22 items, in which each statement is scored by the caregiver using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Total score derived from sub-scores; total ranged from 0-88. Higher scores indicate greater burden. Change: mean score at Week 12 LOCF minus mean score at baseline. Values at final evaluation were imputed using a Last Observation Carried Forward (LOCF) method.
Time Frame: Baseline and Week 12
Population: Per Protocol Set (PPS) was defined as those participants who complied with the study protocol.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Number analyzed (Participants) | 33 | 31 | 33 | 30
Score on a scale
  Baseline | 28.3 (14.4) | 23.2 (11.6) | 26.9 (16.3) | 22.3 (9.8)
  Change from Baseline (LOCF) | -1.3 (11.1) | -0.6 (16.4) | -5.2 (13.8) | 2.9 (9.1)

ADVERSE EVENTS:
Description: Safety Analysis Set (SAS) was defined as all participants who received at least one dose of study drug and had at least one post-baseline safety evaluation.
Arm/Group | 3 mg Donepezil Hydrochloride | 5 mg Donepezil Hydrochloride | 10 mg Donepezil Hydrochloride | Placebo
Serious Adverse Events (participants affected / at risk) | 2/35 | 2/33 | 4/37 | 2/34
Other Adverse Events (participants affected / at risk) | 24/35 | 27/33 | 32/37 | 24/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg Donepezil Hydrochloride (N=35) | 5 mg Donepezil Hydrochloride (N=33) | 10 mg Donepezil Hydrochloride (N=37) | Placebo (N=34)
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 3 mg Donepezil Hydrochloride (N=35) | 5 mg Donepezil Hydrochloride (N=33) | 10 mg Donepezil Hydrochloride (N=37) | Placebo (N=34)
Nasopharyngitis (Infections and infestations) | 3 | 2 | 4 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 3 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Poriomania (Psychiatric disorders) | 2 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 1
Dental Caries (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 0 | 2 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 5 | 3 | 5 | 2
Blood Pressure Increased (Investigations) | 5 | 2 | 2 | 1
Blood Urine Present (Investigations) | 0 | 2 | 4 | 3
Blood Triglycerides Increased (Investigations) | 2 | 1 | 0 | 3
Glucose Urine Present (Investigations) | 0 | 1 | 3 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 4 | 1
Blood Urea Increased (Investigations) | 1 | 0 | 1 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 3
Electrocardiogram QT Prolonged (Investigations) | 0 | 1 | 0 | 2
Protein Urine Present (Investigations) | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No